CLINICAL TRIAL: NCT02632760
Title: Intravenous Iron for Treatment of Anaemia Before Cardiac Surgery
Acronym: ITACS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: National Health and Medical Research Council, Australia (Other); Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 605/15
Record Dates: First submitted 2015-12-07; First posted 2015-12-17 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2024-12

CONDITIONS: Anaemia
MeSH Terms: conditions — Anemia | interventions — ferric carboxymaltose; iron isomaltoside 1000

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ferric carboxymaltose (Active Comparator): ferric carboxymaltose 1000 mg or Iron isomaltoside 1000 mg given Intravenously
  Interventions: Drug: Ferric carboxymaltose
- Placebo (Placebo Comparator): Placebo intravenous infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ferric carboxymaltose — treatment for Iron deficient anaemia
  Other Names: ferinject; Iron isomaltoside
  Arms: ferric carboxymaltose
Drug: Placebo — placebo - no active drug
  Other Names: No active drug
  Arms: Placebo

SUMMARY:
This randomised double-blind, controlled phase IV trial will compare the efficacy, safety and cost-effectiveness of preoperative IV iron with placebo in patients with anaemia before elective cardiac surgery.

DETAILED DESCRIPTION:
Preoperative anaemia is common (≈30%) in patients awaiting cardiac surgery, and is associated with increased complications, ICU and hospital stay, and mortality. The extent of anaemia is worsened by haemodilution occurring with cardiopulmonary bypass and surgical bleeding (average blood loss 0.5-1.5 litres), which in turn impair end-organ blood flow and tissue oxygen delivery. Further, the need for blood transfusion is greatly increased in anaemic patients, and is associated with poor outcomes. In addition, blood transfusions are costly (>$700 per unit), with around 50% of all transfusions used in surgery being for cardiac surgery. The investigators have identified high rates of bleeding complications and transfusion requirements in Australian cardiac surgery; and in another international collaboration, it was found that anaemia, transfusion and kidney injury are inter-related after cardiac surgery. After risk-adjustment, the combination of these three risk factors was associated with a 3.5-fold (95% CI 2.3-5.2) increased odds of kidney injury.

Both anaemia and red cell transfusion are independent risk factors in major surgery. Some of the investigators reviewed Australian cardiac surgery patients from six Victorian hospitals, 2005-2011. We linked the ANZ Society of Cardiothoracic Surgeons cardiac surgery database to laboratory data, including preoperative haemoglobin and all issued blood products (manuscript in preparation). Anaemia was defined according to the WHO definition (Hb <130 g/L for males and <120 g/L for females). There were 15,948 cardiac surgery patients available for inclusion in the analysis, of which 28% were anaemic. Anaemic patients were more likely to receive a red cell transfusion (71% vs. 40%, p<0.001), more transfused units of blood (median 4 [IQR 2-8] vs. 3 [2-5], p<0.001), and had higher 30-day mortality (5.4% vs. 1.9%, p<0.001), new renal failure (43% vs. 26%, p<0.001), and longer hospital stay in survivors (13 days [8-23] vs. 8 days [6-14], p<0.001). After multivariable adjustment, preoperative anaemia was an independent predictor of mortality (adj. OR 1.46, 95% CI 1.14-1.88, p=0.003). Similar results were obtained when restricted to elective surgery, but with hospital stay 9 days (7-17) vs. 7 days (6-11), p<0.001. Other large studies are consistent with this.

The investigators have also analysed data for patients undergoing major non-cardiac surgery from the American College of Surgeons' National Surgical Quality Improvement Program database (a validated outcomes registry from 211 hospitals worldwide). In 227,425 patients undergoing noncardiac surgery, and found that preoperative anaemia was associated with increased 30-day mortality (adj. OR 1.42, 95% CI 1.31-1.54) and morbidity (adj. OR 1.35, 1.30-1.40).

Alfred hospital (Melbourne) transfusion data for 2012-14 (n=2,091) show that anaemic (27% of cohort) and non-anaemic cardiac surgical patients had intraoperative red cell transfusion rates of 31% and 14%, respectively; p<0.01.

Iron deficiency is the commonest cause of anaemia worldwide, and iron deficiency per se independently worsens outcomes after surgery. The traditional textbook definition of iron deficiency anaemia refers to depletion of the body's iron stores due to dietary deficiency or chronic blood loss - an absolute iron deficiency. Chronic disease and inflammation have a direct effect in the pathway of iron absorption and metabolism leading to a state of functional iron deficiency and anaemia. Specifically, the iron regulatory protein hepcidin is upregulated, blocking pathways of iron transport. This prevents iron absorption from the gut, further uptake by the reticuloendothelial system increases stores (ferritin), but distribution and transfer to the bone marrow is blocked. Consequently, despite normal or even increased body iron stores (with normal ferritin levels), these are artifactual, and a state of 'functional iron deficiency' exists. This is commonly seen in renal and cardiac disease and increasingly recognised as a cause for anaemia in the surgical patient. Importantly, IV iron has been shown to overcome this functional deficiency and correct anaemia.

IV iron therapy is effective in treating anaemia in medical (heart failure, kidney disease), post-partum, and preoperative settings (orthopaedic surgery, colon cancer resection, hysterectomy, hip/knee joint replacement. Earlier IV iron preparations using high molecular weight dextran were associated with anaphylaxis due to pre-formed antibodies, but newer preparations are safer, enabling delivery of a full treatment dose in 15 mins, so iron can be administered safely and quickly in outpatients. It is now readily available in Australia and is PBS-listed. This gives patients the equivalent dose of 12 months of tablets in only 15 mins.

Iron deficiency is very common in patients having coronary artery surgery. It is highly plausible that anaemia correction will improve patient outcome following cardiac surgery.However, some data suggest that free iron mediates free radical production associated with organ damage or infection in surgery and this balance between effective anaemia correction and potential risk needs further research. A definitive large trial is needed to determine if IV iron safely, effectively, and promptly corrects preoperative anaemia, and thus reduces risk in cardiac surgery.

The investigators undertook a Cochrane review of iron therapy to treat anaemia in adults including 4,745 participants in 21 trials. This found a trend for better haemoglobin levels with IV iron (MD 0.50 g/dL, 95% CI 0.73-0.27; six studies, N=769) but with considerable, unexplained heterogeneity. Differences in the proportion of participants requiring transfusion were imprecise (RR 0.84, 95% CI 0.66-1.06; 8 studies, N=1,315). Thus the current evidence base is sparse; few randomised trials have been done and these were too small - there remains considerable equipoise.

Review of the literature on anaemia and iron therapy in cardiac surgery, which included 4 small trials of IV iron. Overall, half of all cardiac surgery patients were anaemic before surgery. Preoperative anaemia was found to be independently associated with higher mortality and blood transfusion rate, as well as longer ICU and hospital stay. As also shown by others, preoperative haematocrit was a powerful independent predictor of mortality, renal failure and deep sternal wound infection. In adjusted analyses each 5 point decrease in preoperative haematocrit was associated with an 8% increased risk of death (OR, 1.08; p<0.0003), a 22% increased risk of postoperative renal failure (OR, 1.22; p<0.0001), and a 10% increased risk of deep sternal wound infection (OR, 1.10; p<0.01). There is a need for a well-designed, pragmatic trial to assess the role of preoperative anaemia treatment using IV iron in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with anaemia (males Hb <130 g/L, females <120 g/L) undergoing elective cardiac surgery, and available to receive trial drug 1- 10 weeks prior to surgery

Exclusion Criteria:

* Pregnancy
* Known hypersensitivity to study drug (ferric carboxymaltose or equivalent) or its excipients
* Known or suspected haemoglobinopathy/thalassaemia
* Bone marrow disease
* Haemochromatosis
* Renal dialysis
* Erythropoietin or IV iron in the previous 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 955 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Days alive and out of hospital. | induction of anaesthesia for cardiac surgery up to 90 days post operatively
  90 days post surgery. the number of days the patient was not in hospital or care facility during the 90 day period from surgery.

SECONDARY OUTCOMES:
Correction of anemia following administration of trial drug to day of surgery measure by hemoglobin | from administration of trial drug up to induction of anaesthesia for cardiac surgery up to 10 weeks
  following administration of trial drug to day of surgery. Analysis of the Haemoglobin changes.
Intensive care stay | induction of anaesthesia for cardiac surgery to 30 days post operatively
  Total days in hospital and Intensive care from induction of anaesthesia for cardiac surgery up until 30 days post operation
hospital stay | induction of anaesthesia for cardiac surgery to 30 days post operatively
  Total days in hospital from induction of anaesthesia for cardiac surgery up until 30 days post operation
Disability-free survival | 180 days from induction of anaesthesia for cardiac surgery
  Using the WHODAS to measure disability post operatively up to180 days from surgery. disability will be measured as an increased score of ≥4 for a period of ≥ 3months
90-day survival | induction of anaesthesia for cardiac surgery up to 90 days post operatively
  mortality within 90 days from induction of anaesthesia for cardiac surgery
units of allogeneic blood transfused | induction of anaesthesia for cardiac surgery to discharge from hospital up to 30 days
  number of blood products transfused
person's wellbeing | induction of anaesthesia for cardiac surgery up to 180 days post operatively
  Quality of life after cardiac surgery
Cost-effectiveness | From trial drug administration to 180 days from induction of anaesthesia for cardiac surgery
  comparative cost analysis for the use of iron v's placebo
Days alive and out of hospital. | induction of anaesthesia for cardiac surgery up to 30 days post operatively
  30 days post surgery. the number of days the patient was not in hospital or care facility during the 30 day period from surgery.

OTHER OUTCOMES:
Anaphylaxis | during administration of the trial drug (up to 1 hour)
  drug or transfusion reaction
Infection | induction of anaesthesia for cardiac surgery to 30 days post operatively
  Surgical site infection rate following induction of anaesthesia for cardiac surgery to 30 days post operative

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Myles, MD, Study Chair — Bayside Health
Locations (1):
- Alfred Health, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cameron MJ, Al Kharusi L, Gosselin A, Baradari PG, Chirico A, Amar-Zifkin A, Yang SS. Iron supplementation for patients undergoing cardiac surgery: a protocol for a systematic review and meta-analysis of randomized controlled trials. CMAJ Open. 2021 Jun 4;9(2):E623-E626. doi: 10.9778/cmajo.20200204. Print 2021 Apr-Jun. PMID 34088733
- See also: ITACS web site — https://www.itacs.org.au/